CLINICAL TRIAL: NCT03347396
Title: A Phase 3, Pivotal, Open-label, Multicenter Study to Assess the Efficacy and Safety of Sutimlimab in Patients With Primary Cold Agglutinin Disease Who Have a Recent History of Blood Transfusion
Brief Title: A Study to Assess the Efficacy and Safety of BIVV009 (Sutimlimab) in Participants With Primary Cold Agglutinin Disease Who Have a Recent History of Blood Transfusion (Cardinal Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC16215; BIVV009-03 (Other: Bioverativ Therapeutics Inc.); 2017-003538-10 (EudraCT Number)
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Agglutinin Disease, Cold
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — sutimlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BIVV009 (Experimental): Participants with primary CAD who had a recent history of transfusion (defined as at least 1 transfusion during the last 6 months prior to screening) received an intravenous (IV) infusion of BIVV009 6.5 grams (g) (if body weight was less than [<] 75 kilograms [kg]) or BIVV009 7.5 g (if body weight was greater than or equal to [>=] 75 kg) on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 in Part B, every 2 weeks starting at Week 27 for up to an additional 149 weeks. All participants who completed Part A elected to continue in Part B.
  Interventions: Drug: BIVV009

INTERVENTIONS:
Drug: BIVV009 — Sutimlimab was administered as intravenous (IV) infusion.
  Other Names: Sutimlimab

SUMMARY:
The purpose of Part A was to determine whether sutimlimab administration resulted in a greater than or equal to (>=) 2 grams per deciliter (g/dL) increase in hemoglobin (Hgb) levels or increased Hgb to >= 12 g/dL and obviated the need for blood transfusion during treatment in participants with primary cold agglutinin disease (CAD) who had a recent history of blood transfusion. The purpose of Part B was to evaluate the long-term safety and tolerability of sutimlimab in participants with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of >= 39 kg at screening.
* Confirmed diagnosis of primary CAD based on the following criteria: a) Chronic hemolysis; b) Polyspecific direct antiglobulin test (DAT) positive; c) Monospecific DAT strongly positive for C3d; d) Cold agglutinin titer >= 64 at 4 degree celsius; e) Immunoglobulin G (IgG) DAT less than or equal to (<=) 1+, and f) No overt malignant disease.
* History of at least one documented blood transfusion within 6 months of enrollment.
* Hemoglobin level <= 10.0 g/dL.
* Bilirubin level above the normal reference range, including participants with Gilbert's Syndrome.

Exclusion Criteria:

* Cold agglutinin syndrome secondary to infection, rheumatologic disease, or active hematologic malignancy.
* Clinically relevant infection of any kind within the month preceding enrollment (e.g., active hepatitis C, pneumonia).
* Clinical diagnosis of systemic lupus erythematosus; or other autoimmune disorders with anti-nuclear antibodies at Screening. Anti-nuclear antibodies of long-standing duration without associated clinical symptoms adjudicated on a case-by-case basis during the Confirmatory Review of Patient Eligibility.
* Positive hepatitis panel (including hepatitis B surface antigen and/or hepatitis C virus antibody) prior to or at Screening.
* Positive human immunodeficiency virus (HIV) antibody at screening.
* Treatment with rituximab monotherapy within 3 months or rituximab combination therapies (e.g., with bendamustine, fludarabine, ibrutinib, or cytotoxic drugs) within 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (49):
- United States (13):
  - Arizona Oncology Associates PC, Tucson, Arizona
  - USC/Keck School of Medicine, Los Angeles, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Georgetown University Medical Center, Georgetown, District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Montefiore Medical Center, New York, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UW Hospitals and Clinics, Madison, Wisconsin
- Australia (3):
  - USC Health Clinics, Buderim, Queensland
  - Ballarat Oncology & Haematology, Ballarat, Victoria
  - Monash Medical Centre, Clayton, Victoria
- Medical University of Vienna, Vienna, Austria
- Belgium (3):
  - ZNA Stuivenberg, Antwerp
  - Centre Hospitalier Jolimont, La Louvière
  - University Hospitals Leuven, Leuven
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
  - University of Alberta, Edmonton
- France (3):
  - CHU de Caen, Caen
  - Centre Hospitalier Henri Mondor, Créteil
  - Centre Hospitalier Lyon Sud, Lyon
- Germany (3):
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Universitätsklinikum Essen, Essen
  - Univ Ulm, Inst Klin. Transfusions. Immungen, Ulm
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Laniado Hospital, Netanya
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - A. O. Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - U.O.C. Ematologia- Policlinico "A. Gemelli", Rome
  - U.O.C. Ematologia Ospedale San Bortolo, Vicenza
- Japan (3):
  - Tokai University Hospital, Isehara, Kanagawa
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Juntendo University Nerima Hospital, Tokyo, Tokyo-To
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - St Olavs Hospital, Avdeling for blodsykdommer, Trondheim
- Spain (4):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Clinci i Provincial de Barcelona, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Dr. Peset, Valencia
- United Kingdom (2):
  - St James Hospital, Leeds, Leeds
  - University College London, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Alexander Röth, Wilma Barcellini, Shirley D'Sa, Yoshitaka Miyakawa, Catherine M Broome, Marc Michel, David J. Kuter, Bernd Jilma, Tor Henrik Anderson Tvedt, Stella Lin, Xiaoyu Jiang, Caroline Reuter, William Hobbs, Sigbjørn Berentsen; Inhibition of Complement C1s with Sutimlimab in Patients with Cold Agglutinin Disease (CAD): Results from the Phase 3 Cardinal Study. Blood 2019; 134 (Supplement_2): LBA-2. doi: https://doi.org/10.1182/blood-2019-132490
- [Derived] Roth A, Broome CM, Barcellini W, Tvedt THA, Miyakawa Y, D'Sa S, Cella D, Bozzi S, Jayawardene D, Yoo R, Shafer F, Wardecki M, Weitz IC. Long-term sutimlimab improves quality of life for patients with cold agglutinin disease: CARDINAL 2-year follow-up. Blood Adv. 2023 Oct 10;7(19):5890-5897. doi: 10.1182/bloodadvances.2022009318. PMID 37459203
- [Derived] Roth A, Barcellini W, D'Sa S, Miyakawa Y, Broome CM, Michel M, Kuter DJ, Jilma B, Tvedt THA, Weitz IC, Yoo R, Jayawardene D, Vagge DS, Kralova K, Shafer F, Wardecki M, Lee M, Berentsen S. Sustained inhibition of complement C1s with sutimlimab over 2 years in patients with cold agglutinin disease. Am J Hematol. 2023 Aug;98(8):1246-1253. doi: 10.1002/ajh.26965. Epub 2023 May 29. PMID 37246953
- [Derived] Roth A, Barcellini W, Tvedt THA, Miyakawa Y, Kuter DJ, Su J, Jiang X, Hobbs W, Arias JM, Shafer F, Weitz IC. Sutimlimab improves quality of life in patients with cold agglutinin disease: results of patient-reported outcomes from the CARDINAL study. Ann Hematol. 2022 Oct;101(10):2169-2177. doi: 10.1007/s00277-022-04948-y. Epub 2022 Aug 23. PMID 35999387
- [Derived] Tvedt THA, Steien E, Ovrebo B, Haaverstad R, Hobbs W, Wardecki M, Tjonnfjord GE, Berentsen SA. Sutimlimab, an investigational C1s inhibitor, effectively prevents exacerbation of hemolytic anemia in a patient with cold agglutinin disease undergoing major surgery. Am J Hematol. 2022 Feb 1;97(2):E51-E54. doi: 10.1002/ajh.26409. Epub 2021 Dec 11. No abstract available. PMID 34778998
- [Derived] Roth A, Barcellini W, D'Sa S, Miyakawa Y, Broome CM, Michel M, Kuter DJ, Jilma B, Tvedt THA, Fruebis J, Jiang X, Lin S, Reuter C, Morales-Arias J, Hobbs W, Berentsen S. Sutimlimab in Cold Agglutinin Disease. N Engl J Med. 2021 Apr 8;384(14):1323-1334. doi: 10.1056/NEJMoa2027760. PMID 33826820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 active sites in 8 countries. Out of 42 screened participants, a total of 24 participants were enrolled from 05 March 2018 to 10 Jan 2019. This was a single arm study that consisted of 2 Parts: Part A and Part B.
Pre-assignment Details: Participants were stratified based on baseline body weight to receive BIVV009 6.5 grams (g) (if <75 kg) or 7.5 g (if >=75 kg). As planned, data presented as: 1) Dose-wise (2 dose cohorts: BIVV009 6.5 g & BIVV009 7.5 g) for sections, 'disposition, baseline characteristics, safety endpoints & AEs' and 2) combined population (BIVV009) for efficacy endpoints.
Groups:
- BIVV009 6.5 g: Participants with primary cold agglutinin disease (CAD) and body weight less than (<)75 kg with a recent history of transfusion (defined as at least 1 transfusion during the last 6 months prior to screening in this study) received an intravenous (IV) infusion of BIVV009 6.5 g on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 6.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 143 weeks. All participants who completed Part A elected to continue in Part B.
- BIVV009 7.5 g: Participants with primary CAD and body weight greater than or equal to (>=)75 kg with a recent history of transfusion (defined as at least 1 transfusion during the last 6 months prior to screening in this study) received an IV infusion of BIVV009 7.5 g on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 7.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 149 weeks. All participants who completed Part A elected to continue in Part B.
Period: Part A (26 Weeks)
Arm/Group | BIVV009 6.5 g | BIVV009 7.5 g
Started | 17 | 7
Completed | 16 | 6
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Period: Part B (149 Weeks)
Arm/Group | BIVV009 6.5 g | BIVV009 7.5 g
Started | 16 | 6
Completed | 14 | 5
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- BIVV009 6.5 g: Participants with primary CAD and body weight <75 kg with a recent history of transfusion (defined as at least 1 transfusion during the last 6 months prior to screening in this study) received an IV infusion of BIVV009 6.5 g on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 6.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 143 weeks. All participants who completed Part A elected to continue in Part B.
- BIVV009 7.5 g: Participants with primary CAD and body weight >=75 kg with a recent history of transfusion (defined as at least 1 transfusion during the last 6 months prior to screening in this study) received an IV infusion of BIVV009 7.5 g on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 7.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 149 weeks. All participants who completed Part A elected to continue in Part B.
- Total: Total of all reporting groups
Arm/Group | BIVV009 6.5 g | BIVV009 7.5 g | Total
Number analyzed (Participants) | 17 | 7 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (9.05) | 70.1 (6.01) | 71.3 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants With Response to Treatment
Description: A participant was considered a responder: if he or she did not receive a blood transfusion from Week 5 through Week 26 (end of treatment in Part A) and did not receive treatment for CAD beyond what was permitted per protocol. Additionally, the participant's hemoglobin (Hgb) level must meet either of the following criteria: Hgb level >= 12 grams per deciliter (g/dL) at the treatment assessment endpoint (defined as the average of the values from the Week 23, 25, and 26 visits), or Hgb increased >= 2 g/dL from baseline (defined as the last Hgb value before administration of the first dose of study drug) at treatment assessment endpoint. Percentage of responders was calculated together with a 95% exact Clopper-Pearson confidence interval (CI).
Time Frame: From Week 5 through Week 26
Population: Analysis was performed on Part A-full analysis set (FAS) which included all participants who received at least 1 dose (including partial dose) of study drug. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BIVV009: Participants with primary CAD who had a recent history of blood transfusion (defined as at least 1 transfusion during the last 6 months prior to screening) received an IV infusion of BIVV009 6.5 g (if body weight was <75 kg) or BIVV009 7.5 g (if body weight was >=75 kg) on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 in Part B, every 2 weeks starting at Week 27 for up to an additional 149 weeks. All participants who completed Part A elected to continue in Part B.
Arm/Group | BIVV009
Number analyzed (Participants) | 24
percentage of participants | 54.2 [32.8 to 74.4]

2. Primary Outcome: Part B: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. TESAEs was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the treatment-emergent (TE) period (from the first investigational medicinal product [IMP] administration in Part B to the last IMP administration + 9 weeks follow up period).
Time Frame: Part B, 6.5 g cohort: From first dose (Week 27) up to 143 weeks of treatment + 9 weeks of follow-up (i.e., up to Week 179); Part B, 7.5 g cohort: From first dose (Week 27) up to 149 weeks of treatment + 9 weeks of follow-up (i.e., up to Week 185)
Population: Analysis was performed on Part B safety analysis set (SAS) which included all participants who received at least 1 dose (including partial dose) of study drug in Part B. Data for this outcome measures was planned to be collected and analyzed for dose-wise reporting groups (BIVV009 6.5g and BIVV009 7.5 g).
Measure: Count of Participants; unit: Participants
Groups:
- BIVV009 6.5 g: Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 6.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 143 weeks. All participants who completed Part A elected to continue in Part B.
- BIVV009 7.5 g: Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 7.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 149 weeks. All participants who completed Part A elected to continue in Part B.
Arm/Group | BIVV009 6.5 g | BIVV009 7.5 g
Number analyzed (Participants) | 16 | 6
Participants
  TEAEs | 16 | 6
  TESAEs | 10 | 2

3. Secondary Outcome: Part A: Mean Change From Baseline in Bilirubin Levels at the Treatment Assessment Timepoint
Description: Mean change from baseline in bilirubin levels at the treatment assessment timepoint was reported in this outcome measure. Treatment assessment timepoint was defined as the average of the values from the Week 23, 25, and 26 visits. Least squares (LS) mean and 95% confidence interval (CI) was assessed by Mixed Model for Repeated Measures (MMRM) approach using heterogeneous Toeplitz (TOEPH) covariance matrix with change from baseline as the dependent variable and baseline value and visits as independent variables. Baseline was defined as the last non-missing value prior to the first administration of study drug.
Time Frame: Baseline, treatment assessment timepoint (i.e., average of Week 23, 25 and 26)
Population: Analysis was performed on Part A-FAS. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Least Squares Mean (95% Confidence Interval); unit: micromoles per Liter (mcmol/L)
Arm/Group | BIVV009
Number analyzed (Participants) | 14
micromoles per Liter (mcmol/L) | -38.18 [-42.52 to -33.84]

4. Secondary Outcome: Part A: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score (Quality of Life) at Treatment Assessment Timepoint
Description: FACIT-Fatigue scale consists of 13 questions assessed using a 5-point scale (0=not at all; 1 = a little bit, 2 = somewhat, 3 = quite a bit and 4 = very much). Responses to each question were added to obtain a total score. Total score ranged from 0 to 52, with higher score indicating more fatigue. Treatment assessment timepoint was defined as the average of the values from the Week 23, 25, and 26 visits. LS mean and 95% CI was assessed by MMRM approach using TOEPH covariance matrix with change from baseline as the dependent variable and baseline value and visits as independent variables. Baseline was defined as the last non-missing value prior to the first administration of study drug.
Time Frame: Baseline, treatment assessment timepoint (i.e., average of Week 23, 25 and 26)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BIVV009
Number analyzed (Participants) | 17
score on a scale | 10.85 [8.00 to 13.70]

5. Secondary Outcome: Part A: Mean Change From Baseline in Lactate Dehydrogenase (LDH) at the Treatment Assessment Timepoint
Description: Mean change from baseline in LDH at the treatment assessment timepoint is reported in this outcome measure. Treatment assessment timepoint was defined as the average of the values from the Week 23, 25, and 26 visits. LS mean and 95% CI was assessed by MMRM approach using TOEPH covariance matrix with change from baseline as the dependent variable and baseline value and visits as independent variables. Baseline was defined as the last non-missing value prior to the first administration of study drug.
Time Frame: Baseline, treatment assessment timepoint (i.e., average of Week 23, 25 and 26)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units per liter
Arm/Group | BIVV009
Number analyzed (Participants) | 17
units per liter | -126.95 [-218.47 to -35.42]

6. Secondary Outcome: Part A: Number of Blood Transfusions Per Participant
Description: A participant was to receive a transfusion if his or her Hgb level met either of the following criteria: Hgb was <9 g/dL and the participant had symptoms of anemia or Hgb was <7 g/dL and the participant was asymptomatic. Number of transfusions after the first 5 weeks of study drug administration and up to Week 26 are reported in this outcome measure.
Time Frame: From Week 5 up to Week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: blood transfusions per participant
Arm/Group | BIVV009
Number analyzed (Participants) | 23
blood transfusions per participant | 0.9 (2.75)

7. Secondary Outcome: Part A: Number of Blood Units Transfused Per Participant
Description: A participant was to receive a transfusion if his or her Hgb level met either of the following criteria: -Hgb was <9 g/dL and the participant had symptoms of anemia or Hgb was <7 g/dL and the participant was asymptomatic. Number of blood units transfused after the first 5 weeks of study drug administration and up to Week 26 are reported in this outcome measure.
Time Frame: From Week 5 up to Week 26
Population: Analysis was performed on Part A-FAS. Here, 'overall number of participants analyzed' = number of participants with at least 1 transfusion. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: blood units transfused per participant
Arm/Group | BIVV009
Number analyzed (Participants) | 6
blood units transfused per participant | 5.8 (8.47)

8. Secondary Outcome: Part A: Mean Change From Baseline in Hemoglobin (Hgb) Level at the Treatment Assessment Timepoint
Description: Mean change from baseline (Week 0) in Hgb at treatment assessment timepoint is reported in this outcome measure. Treatment assessment timepoint was defined as the average of the values from the Week 23, 25, and 26 visits. LS mean and 95% CI was assessed by MMRM approach using TOEPH covariance matrix with change from baseline as the dependent variable and baseline value and visits as independent variables. Baseline was defined as the last non-missing value prior to the first administration of study drug.
Time Frame: Baseline, treatment assessment timepoint (i.e., average of Week 23, 25 and 26)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | BIVV009
Number analyzed (Participants) | 17
g/dL | 2.60 [0.74 to 4.46]

9. Secondary Outcome: Part B: Change From Baseline in Hemoglobin (Hgb) Level at Each Specified Time Points
Description: Change From Hgb level from baseline (Week 0) at each specified time points (i.e., Weeks 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65, 67, 69, 71, 73, 75, 77, 79, 83, 87, 91, 95, 99, 103, 107, 111, 115, 119, 123, 127, 131, 135, 139, 143, 147, 151, 155, 159, 163, 167, 171, 175 and early termination/safety follow up [ET/SFU] Visit) is reported in this outcome measure. Baseline was defined as the last non-missing value prior to the first administration of study drug in Part A. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 185).
Time Frame: Baseline, Weeks 27,29,31,33,35,37,39,41, 43, 45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65, 67, 69, 71, 73, 75, 77, 79, 83, 87, 91, 95, 99, 103, 107, 111, 115, 119, 123, 127, 131, 135, 139, 143, 147, 151, 155, 159, 163, 167, 171, 175, ET/SFU (up to Week 185)
Population: Analysis was performed on Part B-FAS which included all participants who enrolled in Part B study and received at least 1 dose (including partial dose) of study drug. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | BIVV009
Number analyzed (Participants) | 22
g/dL
  Week 27 | 2.76 (2.20)
  Week 29 | 2.77 (2.20)
  Week 31 | 2.74 (1.96)
  Week 33 | 2.87 (1.97)
  Week 35: number analyzed (Participants) | 21
  Week 35 | 2.82 (2.10)
  Week 37: number analyzed (Participants) | 21
  Week 37 | 2.71 (2.08)
  Week 39: number analyzed (Participants) | 21
  Week 39 | 2.72 (2.26)
  Week 41: number analyzed (Participants) | 21
  Week 41 | 2.76 (2.24)
  Week 43: number analyzed (Participants) | 21
  Week 43 | 2.73 (2.06)
  Week 45: number analyzed (Participants) | 21
  Week 45 | 2.84 (2.21)
  Week 47: number analyzed (Participants) | 21
  Week 47 | 2.74 (1.95)
  Week 49: number analyzed (Participants) | 21
  Week 49 | 2.73 (2.09)
  Week 51 | 2.71 (1.97)
  Week 53 | 2.66 (1.97)
  Week 55: number analyzed (Participants) | 21
  Week 55 | 2.73 (1.96)
  Week 57: number analyzed (Participants) | 21
  Week 57 | 3.01 (2.36)
  Week 59: number analyzed (Participants) | 21
  Week 59 | 2.81 (2.10)
  Week 61: number analyzed (Participants) | 21
  Week 61 | 2.88 (2.37)
  Week 63: number analyzed (Participants) | 21
  Week 63 | 2.99 (2.33)
  Week 65: number analyzed (Participants) | 21
  Week 65 | 2.53 (2.18)
  Week 67: number analyzed (Participants) | 20
  Week 67 | 2.52 (2.20)
  Week 69: number analyzed (Participants) | 20
  Week 69 | 2.96 (2.08)
  Week 71: number analyzed (Participants) | 19
  Week 71 | 2.86 (2.31)
  Week 73: number analyzed (Participants) | 20
  Week 73 | 2.79 (2.25)
  Week 75: number analyzed (Participants) | 21
  Week 75 | 2.70 (2.18)
  Week 77: number analyzed (Participants) | 21
  Week 77 | 2.93 (2.59)
  Week 79: number analyzed (Participants) | 19
  Week 79 | 3.13 (2.23)
  Week 83: number analyzed (Participants) | 20
  Week 83 | 2.89 (2.47)
  Week 87: number analyzed (Participants) | 18
  Week 87 | 2.63 (2.36)
  Week 91: number analyzed (Participants) | 20
  Week 91 | 3.23 (2.17)
  Week 95: number analyzed (Participants) | 19
  Week 95 | 3.12 (2.06)
  Week 99: number analyzed (Participants) | 20
  Week 99 | 2.98 (2.01)
  Week 103: number analyzed (Participants) | 21
  Week 103 | 2.92 (2.09)
  Week 107: number analyzed (Participants) | 21
  Week 107 | 2.60 (2.10)
  Week 111: number analyzed (Participants) | 21
  Week 111 | 2.82 (2.17)
  Week 115: number analyzed (Participants) | 19
  Week 115 | 2.96 (2.25)
  Week 119: number analyzed (Participants) | 20
  Week 119 | 2.79 (2.57)
  Week 123: number analyzed (Participants) | 20
  Week 123 | 2.82 (2.35)
  Week 127: number analyzed (Participants) | 19
  Week 127 | 2.89 (1.99)
  Week 131: number analyzed (Participants) | 19
  Week 131 | 3.03 (2.19)
  Week 135: number analyzed (Participants) | 19
  Week 135 | 3.35 (1.99)
  Week 139: number analyzed (Participants) | 13
  Week 139 | 3.42 (2.14)
  Week 143: number analyzed (Participants) | 11
  Week 143 | 3.43 (2.31)
  Week 147: number analyzed (Participants) | 8
  Week 147 | 3.75 (2.38)
  Week 151: number analyzed (Participants) | 8
  Week 151 | 3.43 (1.91)
  Week 155: number analyzed (Participants) | 8
  Week 155 | 3.74 (1.94)
  Week 159: number analyzed (Participants) | 6
  Week 159 | 5.20 (1.65)
  Week 163: number analyzed (Participants) | 4
  Week 163 | 4.18 (1.14)
  Week 167: number analyzed (Participants) | 2
  Week 167 | 4.80 (0.42)
  Week 171: number analyzed (Participants) | 1
  Week 171 | 4.80
  Week 175: number analyzed (Participants) | 1
  Week 175 | 4.40
  ET/SFU Visit: number analyzed (Participants) | 20
  ET/SFU Visit | 1.21 (1.56)

10. Secondary Outcome: Part B: Change From Baseline in Bilirubin Levels at Each Specified Time Points
Description: Change from baseline (Week 0) in bilirubin levels at each specified time point (i.e., Weeks 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65, 67, 69, 71, 73, 75, 77, 79, 83, 87, 91, 95, 99, 103, 107, 111, 115, 119, 123, 127, 131, 135, 139, 143, 147, 151, 155, 159, 163, 167, 171, 175 and ET/SFU Visit) is reported in this outcome measure. Baseline was defined as the last non-missing value prior to the first administration of study drug in Part A. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 185).
Time Frame: as for outcome 9
Population: Analysis was performed on Part B-FAS. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | BIVV009
Number analyzed (Participants) | 19
mcmol/L
  Week 27 | -34.96 (18.31)
  Week 29 | -34.92 (15.78)
  Week 31 | -32.58 (17.07)
  Week 33 | -32.67 (17.52)
  Week 35 | -32.25 (22.39)
  Week 37 | -33.24 (15.53)
  Week 39: number analyzed (Participants) | 13
  Week 39 | -35.92 (13.17)
  Week 41: number analyzed (Participants) | 18
  Week 41 | -35.03 (13.71)
  Week 43: number analyzed (Participants) | 16
  Week 43 | -36.46 (17.25)
  Week 45: number analyzed (Participants) | 18
  Week 45 | -34.81 (15.76)
  Week 47: number analyzed (Participants) | 18
  Week 47 | -34.57 (16.53)
  Week 49: number analyzed (Participants) | 18
  Week 49 | -32.36 (19.50)
  Week 51: number analyzed (Participants) | 16
  Week 51 | -34.88 (15.90)
  Week 53 | -35.25 (18.32)
  Week 55: number analyzed (Participants) | 18
  Week 55 | -34.79 (16.70)
  Week 57: number analyzed (Participants) | 18
  Week 57 | -36.32 (16.54)
  Week 59: number analyzed (Participants) | 18
  Week 59 | -35.77 (17.73)
  Week 61: number analyzed (Participants) | 18
  Week 61 | -36.39 (16.14)
  Week 63: number analyzed (Participants) | 17
  Week 63 | -38.25 (15.43)
  Week 65: number analyzed (Participants) | 17
  Week 65 | -35.46 (16.84)
  Week 67: number analyzed (Participants) | 17
  Week 67 | -35.74 (18.37)
  Week 69: number analyzed (Participants) | 17
  Week 69 | -33.88 (16.83)
  Week 71: number analyzed (Participants) | 17
  Week 71 | -32.54 (23.01)
  Week 73: number analyzed (Participants) | 14
  Week 73 | -33.03 (21.82)
  Week 75: number analyzed (Participants) | 16
  Week 75 | -30.55 (21.68)
  Week 77: number analyzed (Participants) | 18
  Week 77 | -30.95 (22.83)
  Week 79: number analyzed (Participants) | 17
  Week 79 | -35.51 (14.79)
  Week 83: number analyzed (Participants) | 16
  Week 83 | -38.60 (13.90)
  Week 87: number analyzed (Participants) | 15
  Week 87 | -37.45 (16.29)
  Week 91: number analyzed (Participants) | 16
  Week 91 | -35.19 (16.07)
  Week 95: number analyzed (Participants) | 15
  Week 95 | -33.57 (15.93)
  Week 99: number analyzed (Participants) | 15
  Week 99 | -28.71 (21.98)
  Week 103: number analyzed (Participants) | 18
  Week 103 | -32.04 (22.45)
  Week 107: number analyzed (Participants) | 18
  Week 107 | -34.46 (15.27)
  Week 111: number analyzed (Participants) | 15
  Week 111 | -37.67 (14.28)
  Week 115: number analyzed (Participants) | 16
  Week 115 | -36.41 (16.76)
  Week 119: number analyzed (Participants) | 16
  Week 119 | -34.65 (13.71)
  Week 123: number analyzed (Participants) | 17
  Week 123 | -29.99 (24.96)
  Week 127: number analyzed (Participants) | 17
  Week 127 | -35.57 (17.83)
  Week 131: number analyzed (Participants) | 16
  Week 131 | -35.03 (18.72)
  Week 135: number analyzed (Participants) | 15
  Week 135 | -36.88 (14.71)
  Week 139: number analyzed (Participants) | 11
  Week 139 | -37.60 (14.59)
  Week 143: number analyzed (Participants) | 8
  Week 143 | -44.50 (15.96)
  Week 147: number analyzed (Participants) | 6
  Week 147 | -44.82 (15.12)
  Week 151: number analyzed (Participants) | 6
  Week 151 | -46.53 (10.80)
  Week 155: number analyzed (Participants) | 6
  Week 155 | -50.32 (12.63)
  Week 159: number analyzed (Participants) | 5
  Week 159 | -46.30 (13.90)
  Week 163: number analyzed (Participants) | 4
  Week 163 | -46.13 (11.86)
  Week 167: number analyzed (Participants) | 2
  Week 167 | -36.30 (12.59)
  Week 171: number analyzed (Participants) | 1
  Week 171 | -32.50
  Week 175: number analyzed (Participants) | 1
  Week 175 | -29.10
  ET/SFU Visit: number analyzed (Participants) | 17
  ET/SFU Visit | -9.98 (18.11)

11. Secondary Outcome: Part B: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score (Quality of Life) at Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135, 147,159, 171 and Early Termination (ET) Visit/Safety Follow-up Visit
Description: FACIT-Fatigue scale consists of 13 questions assessed using a 5-point scale (0=not at all; 1 = a little bit, 2 = somewhat, 3 = quite a bit and 4 = very much). Responses to each question were added to obtain a total score. The Total score ranged from 0 to 52, with higher score indicating more fatigue. Baseline (Week 0) was defined as the last non-missing value prior to the first administration of study drug in Part A. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 185).
Time Frame: Baseline, Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135, 147,159, 171 and ET Visit/SFU visit (i.e., up to Week 185)
Population: Analysis was performed on Part B-FAS. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV009
Number analyzed (Participants) | 22
score on a scale
  Week 39: number analyzed (Participants) | 19
  Week 39 | 9.37 (16.00)
  Week 51: number analyzed (Participants) | 20
  Week 51 | 10.50 (12.05)
  Week 63: number analyzed (Participants) | 19
  Week 63 | 10.21 (11.88)
  Week 75: number analyzed (Participants) | 19
  Week 75 | 11.00 (11.51)
  Week 87: number analyzed (Participants) | 18
  Week 87 | 10.39 (13.41)
  Week 99: number analyzed (Participants) | 17
  Week 99 | 9.94 (8.19)
  Week 111: number analyzed (Participants) | 18
  Week 111 | 9.11 (12.35)
  Week 123: number analyzed (Participants) | 19
  Week 123 | 6.79 (11.28)
  Week 135: number analyzed (Participants) | 14
  Week 135 | 11.71 (13.85)
  Week 147: number analyzed (Participants) | 7
  Week 147 | 13.29 (13.39)
  Week 159: number analyzed (Participants) | 4
  Week 159 | 24.75 (10.24)
  Week 171: number analyzed (Participants) | 1
  Week 171 | 32.00
  ET/SFU Visit: number analyzed (Participants) | 19
  ET/SFU Visit | 1.05 (8.15)

12. Secondary Outcome: Part B: Change From Baseline in 12-Item Short-Form Survey (SF-12) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores at Each Specified Time Points
Description: SF-12: 12 item-questionnaire assessed health-related quality of life (HRQOL) contained 12 items, categorized into 8 domains (subscales) of functioning and well-being: physical functioning, role-physical, role emotional, mental health, bodily pain, general health, vitality and social functioning, with each domain score ranged from 0 (poor health) to 100 (better health). Higher scores = good health condition. These 8 domains were further summarized into 2 summary scores, PCS and MCS for which, score ranged 0 (poor health) to 100 (better health). Higher scores = better HRQOL. Baseline (Week 0) was defined as the last non-missing value prior to first administration of study drug in Part A. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 185). Change from baseline in SF-12 PCS and MCS scores is reported in this outcome measure.
Time Frame: Baseline, Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135 and ET Visit/SFU visit (i.e., up to Week 185)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV009
Number analyzed (Participants) | 22
score on a scale
  Week 39-PCS: number analyzed (Participants) | 16
  Week 39-PCS | 7.813 (10.486)
  Week 39-MCS: number analyzed (Participants) | 16
  Week 39-MCS | 5.859 (10.249)
  Week 51-PCS: number analyzed (Participants) | 18
  Week 51-PCS | 6.677 (9.925)
  Week 51-MCS: number analyzed (Participants) | 18
  Week 51-MCS | 3.912 (9.493)
  Week 63-PCS: number analyzed (Participants) | 19
  Week 63-PCS | 8.318 (7.148)
  Week 63-MCS: number analyzed (Participants) | 19
  Week 63-MCS | 2.385 (9.777)
  Week 75-PCS: number analyzed (Participants) | 18
  Week 75-PCS | 6.580 (9.214)
  Week 75-MCS: number analyzed (Participants) | 18
  Week 75-MCS | 3.102 (9.881)
  Week 87-PCS: number analyzed (Participants) | 18
  Week 87-PCS | 6.398 (9.021)
  Week 87-MCS: number analyzed (Participants) | 18
  Week 87-MCS | 1.611 (10.336)
  Week 99-PCS: number analyzed (Participants) | 14
  Week 99-PCS | 9.054 (5.803)
  Week 99-MCS: number analyzed (Participants) | 14
  Week 99-MCS | 2.581 (9.169)
  Week 111-PCS: number analyzed (Participants) | 8
  Week 111-PCS | 11.958 (3.832)
  Week 111-MCS: number analyzed (Participants) | 8
  Week 111-MCS | 2.523 (12.585)
  Week 123-PCS: number analyzed (Participants) | 6
  Week 123-PCS | 4.743 (6.900)
  Week 123-MCS: number analyzed (Participants) | 6
  Week 123-MCS | 3.810 (14.071)
  Week 135-PCS: number analyzed (Participants) | 1
  Week 135-PCS | 10.450
  Week 135-MCS: number analyzed (Participants) | 1
  Week 135-MCS | 27.900
  ET/SFU Visit-PCS: number analyzed (Participants) | 1
  ET/SFU Visit-PCS | -8.920
  ET/SFU Visit-MCS: number analyzed (Participants) | 1
  ET/SFU Visit-MCS | -1.180

13. Secondary Outcome: Part B: Change From Baseline in 5-level European Quality of Life 5-Dimensions 5-Level Questionnaire (EQ-5D-5L) Health State Utility Index and VAS Scores at Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135, 147,159, 171 and ET Visit/SFU Visit
Description: EQ-5D-5L:standardized, participant-rated questionnaire to assess health-related quality of life. EQ-5D-5L includes 2 components: EQ-5D-5L health state utility index (descriptive system) and Visual Analog Scale (VAS). EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response option: no problems, slight problems, moderate problems, severe problems, and extreme problems measured with Likert scale. EQ-5D-5L responses relating to 5 dimensions are converted into a single index utility score between 0 to 1, where higher score=better health state. The EQ-5D-5L VAS rated participant's current health state on a scale from 0=worst imaginable health state to 100 =best imaginable health state. Baseline (Week 0): last non-missing value prior to first administration of study drug in Part A. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 185).
Time Frame: Baseline, Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135, 147,159, 171 and ET Visit/SFU visit (i.e., up to Week 185)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV009
Number analyzed (Participants) | 22
score on a scale
  Week 39 - Index score: number analyzed (Participants) | 18
  Week 39 - Index score | 0.067 (0.264)
  Week 39 - VAS score: number analyzed (Participants) | 18
  Week 39 - VAS score | 18.111 (20.642)
  Week 51 - Index score: number analyzed (Participants) | 20
  Week 51 - Index score | 0.078 (0.194)
  Week 51 - VAS score: number analyzed (Participants) | 20
  Week 51 - VAS score | 14.500 (19.050)
  Week 63 - Index score: number analyzed (Participants) | 19
  Week 63 - Index score | 0.092 (0.166)
  Week 63 - VAS score: number analyzed (Participants) | 19
  Week 63 - VAS score | 18.053 (16.844)
  Week 75 - Index score: number analyzed (Participants) | 19
  Week 75 - Index score | 0.069 (0.211)
  Week 75 - VAS score: number analyzed (Participants) | 19
  Week 75 - VAS score | 17.842 (16.604)
  Week 87 - Index score: number analyzed (Participants) | 19
  Week 87 - Index score | 0.022 (0.226)
  Week 87 - VAS score: number analyzed (Participants) | 19
  Week 87 - VAS score | 14.421 (20.815)
  Week 99 - Index Score: number analyzed (Participants) | 17
  Week 99 - Index Score | 0.060 (0.136)
  Week 99 - VAS Score: number analyzed (Participants) | 17
  Week 99 - VAS Score | 14.059 (13.818)
  Week 111 - Index score: number analyzed (Participants) | 18
  Week 111 - Index score | 0.099 (0.174)
  Week 111 - VAS score: number analyzed (Participants) | 18
  Week 111 - VAS score | 18.889 (15.408)
  Week 123 - Index Score: number analyzed (Participants) | 19
  Week 123 - Index Score | 0.009 (0.190)
  Week 123 - VAS score: number analyzed (Participants) | 19
  Week 123 - VAS score | 8.842 (18.765)
  Week 135 - Index score: number analyzed (Participants) | 15
  Week 135 - Index score | 0.085 (0.233)
  Week 135 - VAS score: number analyzed (Participants) | 15
  Week 135 - VAS score | 17.067 (21.608)
  Week 147 - Index score: number analyzed (Participants) | 7
  Week 147 - Index score | 0.143 (0.131)
  Week 147 - VAS score: number analyzed (Participants) | 7
  Week 147 - VAS score | 17.857 (20.178)
  Week 159 - Index Score: number analyzed (Participants) | 4
  Week 159 - Index Score | 0.250 (0.145)
  Week 159 - VAS score: number analyzed (Participants) | 4
  Week 159 - VAS score | 36.250 (14.930)
  Week 171 - Index score: number analyzed (Participants) | 1
  Week 171 - Index score | 0.535
  Week 171 - VAS score: number analyzed (Participants) | 1
  Week 171 - VAS score | 35.000
  ET/SFU Visit - Index score: number analyzed (Participants) | 19
  ET/SFU Visit - Index score | -0.025 (0.173)
  ET/SFU Visit - VAS score: number analyzed (Participants) | 19
  ET/SFU Visit - VAS score | 1.263 (19.287)

14. Secondary Outcome: Part B: Number of Participants With Response to Participant's Global Impression of (Fatigue) Severity (PGIS) Questionnaire at Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135, 147,159, 171 and at ET Visit/SFU Visit
Description: The PGIS is a self-reported scale. The PGIS is a 1-item questionnaire designed to assess participant's impression of disease severity using a 5-point scale ranging from 1 to 5, where 1=none, 2= mild, 3=moderate, 4=severe, 5=very severe. Higher scores indicated greater severity. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 185).
Time Frame: At Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135, 147,159, 171 and at ET Visit/SFU visit (i.e., up to Week 185)
Population: Analysis was performed on Part B-FAS population. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Count of Participants; unit: Participants
Arm/Group | BIVV009
Number analyzed (Participants) | 22
Participants
  Week 39 - None: number analyzed (Participants) | 18
  Week 39 - None | 5
  Week 39 - Mild: number analyzed (Participants) | 18
  Week 39 - Mild | 8
  Week 39 - Moderate: number analyzed (Participants) | 18
  Week 39 - Moderate | 4
  Week 39 - Severe: number analyzed (Participants) | 18
  Week 39 - Severe | 1
  Week 39 - Very severe: number analyzed (Participants) | 18
  Week 39 - Very severe | 0
  Week 51 - None: number analyzed (Participants) | 21
  Week 51 - None | 5
  Week 51 - Mild: number analyzed (Participants) | 21
  Week 51 - Mild | 13
  Week 51 - Moderate: number analyzed (Participants) | 21
  Week 51 - Moderate | 3
  Week 51 - Severe: number analyzed (Participants) | 21
  Week 51 - Severe | 0
  Week 51 - Very severe: number analyzed (Participants) | 21
  Week 51 - Very severe | 0
  Week 63 - None: number analyzed (Participants) | 20
  Week 63 - None | 4
  Week 63 - Mild: number analyzed (Participants) | 20
  Week 63 - Mild | 12
  Week 63 - Moderate: number analyzed (Participants) | 20
  Week 63 - Moderate | 3
  Week 63 - Severe: number analyzed (Participants) | 20
  Week 63 - Severe | 1
  Week 63 - Very severe: number analyzed (Participants) | 20
  Week 63 - Very severe | 0
  Week 75 - None: number analyzed (Participants) | 20
  Week 75 - None | 3
  Week 75 - Mild: number analyzed (Participants) | 20
  Week 75 - Mild | 12
  Week 75 - Moderate: number analyzed (Participants) | 20
  Week 75 - Moderate | 5
  Week 75 - Severe: number analyzed (Participants) | 20
  Week 75 - Severe | 0
  Week 75 - Very severe: number analyzed (Participants) | 20
  Week 75 - Very severe | 0
  Week 87 - None: number analyzed (Participants) | 19
  Week 87 - None | 5
  Week 87 - Mild: number analyzed (Participants) | 19
  Week 87 - Mild | 9
  Week 87 - Moderate: number analyzed (Participants) | 19
  Week 87 - Moderate | 3
  Week 87 - Severe: number analyzed (Participants) | 19
  Week 87 - Severe | 2
  Week 87 - Very severe: number analyzed (Participants) | 19
  Week 87 - Very severe | 0
  Week 99 - None: number analyzed (Participants) | 18
  Week 99 - None | 4
  Week 99 - Mild: number analyzed (Participants) | 18
  Week 99 - Mild | 10
  Week 99 - Moderate: number analyzed (Participants) | 18
  Week 99 - Moderate | 4
  Week 99 - Severe: number analyzed (Participants) | 18
  Week 99 - Severe | 0
  Week 99 - Very severe: number analyzed (Participants) | 18
  Week 99 - Very severe | 0
  Week 111 - None: number analyzed (Participants) | 19
  Week 111 - None | 7
  Week 111 - Mild: number analyzed (Participants) | 19
  Week 111 - Mild | 6
  Week 111 - Moderate: number analyzed (Participants) | 19
  Week 111 - Moderate | 6
  Week 111 - Severe: number analyzed (Participants) | 19
  Week 111 - Severe | 0
  Week 111 - Very severe: number analyzed (Participants) | 19
  Week 111 - Very severe | 0
  Week 123 - None: number analyzed (Participants) | 20
  Week 123 - None | 4
  Week 123 - Mild: number analyzed (Participants) | 20
  Week 123 - Mild | 7
  Week 123 - Moderate: number analyzed (Participants) | 20
  Week 123 - Moderate | 7
  Week 123 - Severe: number analyzed (Participants) | 20
  Week 123 - Severe | 2
  Week 123 - Very severe: number analyzed (Participants) | 20
  Week 123 - Very severe | 0
  Week 135 - None: number analyzed (Participants) | 15
  Week 135 - None | 4
  Week 135 - Mild: number analyzed (Participants) | 15
  Week 135 - Mild | 8
  Week 135 - Moderate: number analyzed (Participants) | 15
  Week 135 - Moderate | 3
  Week 135 - Severe: number analyzed (Participants) | 15
  Week 135 - Severe | 0
  Week 135 - Very severe: number analyzed (Participants) | 15
  Week 135 - Very severe | 0
  Week 147 - None: number analyzed (Participants) | 7
  Week 147 - None | 3
  Week 147 - Mild: number analyzed (Participants) | 7
  Week 147 - Mild | 3
  Week 147 - Moderate: number analyzed (Participants) | 7
  Week 147 - Moderate | 1
  Week 147 - Severe: number analyzed (Participants) | 7
  Week 147 - Severe | 0
  Week 147 - Very severe: number analyzed (Participants) | 7
  Week 147 - Very severe | 0
  Week 159 - None: number analyzed (Participants) | 4
  Week 159 - None | 3
  Week 159 - Mild: number analyzed (Participants) | 4
  Week 159 - Mild | 1
  Week 159 - Moderate: number analyzed (Participants) | 4
  Week 159 - Moderate | 0
  Week 159 - Severe: number analyzed (Participants) | 4
  Week 159 - Severe | 0
  Week 159 - Very severe: number analyzed (Participants) | 4
  Week 159 - Very severe | 0
  Week 171 - None: number analyzed (Participants) | 1
  Week 171 - None | 0
  Week 171 - Mild: number analyzed (Participants) | 1
  Week 171 - Mild | 1
  Week 171 - Moderate: number analyzed (Participants) | 1
  Week 171 - Moderate | 0
  Week 171 - Severe: number analyzed (Participants) | 1
  Week 171 - Severe | 0
  Week 171 - Very severe: number analyzed (Participants) | 1
  Week 171 - Very severe | 0
  ET/SFU Visit - None: number analyzed (Participants) | 20
  ET/SFU Visit - None | 4
  ET/SFU Visit - Mild: number analyzed (Participants) | 20
  ET/SFU Visit - Mild | 6
  ET/SFU Visit - Moderate: number analyzed (Participants) | 20
  ET/SFU Visit - Moderate | 4
  ET/SFU Visit - Severe: number analyzed (Participants) | 20
  ET/SFU Visit - Severe | 5
  ET/SFU Visit - Very severe: number analyzed (Participants) | 20
  ET/SFU Visit - Very severe | 1

15. Secondary Outcome: Part B: Number of Participants With Response to Participant's Global Impression of Change (PGIC) Questionnaire at Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135, 147,159, 171 and at ET Visit/SFU Visit
Description: PGIC is a self-administered questionnaire to evaluate the improvement or worsening compared to the start of the study. PGIC was assessed on a 7-point Likert scale ranged from 1 (greatly improved) to 7 (greatly worsened). Categories were defined based on the PGIC scores as follows: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse and 7=very much worsen. Higher scores indicated greater severity. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 185).
Time Frame: At Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135, 147,159, 171 and at ET Visit/SFU visit (i.e., up to Week 185)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | BIVV009
Number analyzed (Participants) | 22
Participants
  Week 39 - Very much improved: number analyzed (Participants) | 19
  Week 39 - Very much improved | 9
  Week 39 - Much improved: number analyzed (Participants) | 19
  Week 39 - Much improved | 5
  Week 39 - Minimally improved: number analyzed (Participants) | 19
  Week 39 - Minimally improved | 3
  Week 39 - No change: number analyzed (Participants) | 19
  Week 39 - No change | 1
  Week 39 - Minimally worse: number analyzed (Participants) | 19
  Week 39 - Minimally worse | 0
  Week 39 - Much worse: number analyzed (Participants) | 19
  Week 39 - Much worse | 1
  Week 39 - Very much worse: number analyzed (Participants) | 19
  Week 39 - Very much worse | 0
  Week 51 - Very much improved: number analyzed (Participants) | 21
  Week 51 - Very much improved | 6
  Week 51 - Much improved: number analyzed (Participants) | 21
  Week 51 - Much improved | 13
  Week 51 - Minimally improved: number analyzed (Participants) | 21
  Week 51 - Minimally improved | 2
  Week 51 - No change: number analyzed (Participants) | 21
  Week 51 - No change | 0
  Week 51 - Minimally worse: number analyzed (Participants) | 21
  Week 51 - Minimally worse | 0
  Week 51 - Much worse: number analyzed (Participants) | 21
  Week 51 - Much worse | 0
  Week 51- Very much worse: number analyzed (Participants) | 21
  Week 51- Very much worse | 0
  Week 63 - Very much improved: number analyzed (Participants) | 20
  Week 63 - Very much improved | 8
  Week 63 - Much improved: number analyzed (Participants) | 20
  Week 63 - Much improved | 9
  Week 63 - Minimally improved: number analyzed (Participants) | 20
  Week 63 - Minimally improved | 1
  Week 63 - No change: number analyzed (Participants) | 20
  Week 63 - No change | 1
  Week 63 - Minimally worse: number analyzed (Participants) | 20
  Week 63 - Minimally worse | 1
  Week 63 - Much worse: number analyzed (Participants) | 20
  Week 63 - Much worse | 0
  Week 63 - Very much worse: number analyzed (Participants) | 20
  Week 63 - Very much worse | 0
  Week 75 - Very much improved: number analyzed (Participants) | 20
  Week 75 - Very much improved | 5
  Week 75 - Much improved: number analyzed (Participants) | 20
  Week 75 - Much improved | 11
  Week 75 - Minimally improved: number analyzed (Participants) | 20
  Week 75 - Minimally improved | 1
  Week 75 - No change: number analyzed (Participants) | 20
  Week 75 - No change | 2
  Week 75 - Minimally worse: number analyzed (Participants) | 20
  Week 75 - Minimally worse | 1
  Week 75 - Much worse: number analyzed (Participants) | 20
  Week 75 - Much worse | 0
  Week 75 - Very much worse: number analyzed (Participants) | 20
  Week 75 - Very much worse | 0
  Week 87 - Very much improved: number analyzed (Participants) | 19
  Week 87 - Very much improved | 5
  Week 87 - Much improved: number analyzed (Participants) | 19
  Week 87 - Much improved | 11
  Week 87 - Minimally improved: number analyzed (Participants) | 19
  Week 87 - Minimally improved | 2
  Week 87 - No change: number analyzed (Participants) | 19
  Week 87 - No change | 1
  Week 87 - Minimally worse: number analyzed (Participants) | 19
  Week 87 - Minimally worse | 0
  Week 87 - Much worse: number analyzed (Participants) | 19
  Week 87 - Much worse | 0
  Week 87 - Very much worse: number analyzed (Participants) | 19
  Week 87 - Very much worse | 0
  Week 99 - Very much improved: number analyzed (Participants) | 18
  Week 99 - Very much improved | 4
  Week 99 - Much improved: number analyzed (Participants) | 18
  Week 99 - Much improved | 10
  Week 99 - Minimally improved: number analyzed (Participants) | 18
  Week 99 - Minimally improved | 3
  Week 99 - No Change: number analyzed (Participants) | 18
  Week 99 - No Change | 1
  Week 99 - Minimally worse: number analyzed (Participants) | 18
  Week 99 - Minimally worse | 0
  Week 99 - Much worse: number analyzed (Participants) | 18
  Week 99 - Much worse | 0
  Week 99 - Very much worse: number analyzed (Participants) | 18
  Week 99 - Very much worse | 0
  Week 111 - Very much improved: number analyzed (Participants) | 19
  Week 111 - Very much improved | 7
  Week 111 - Much improved: number analyzed (Participants) | 19
  Week 111 - Much improved | 7
  Week 111 - Minimally improved: number analyzed (Participants) | 19
  Week 111 - Minimally improved | 5
  Week 111 - No change: number analyzed (Participants) | 19
  Week 111 - No change | 0
  Week 111 - Minimally worse: number analyzed (Participants) | 19
  Week 111 - Minimally worse | 0
  Week 111 - Much worse: number analyzed (Participants) | 19
  Week 111 - Much worse | 0
  Week 111 - Very much worse: number analyzed (Participants) | 19
  Week 111 - Very much worse | 0
  Week 123 - Very much improved: number analyzed (Participants) | 20
  Week 123 - Very much improved | 8
  Week 123 - Much improved: number analyzed (Participants) | 20
  Week 123 - Much improved | 6
  Week 123 - Minimally improved: number analyzed (Participants) | 20
  Week 123 - Minimally improved | 6
  Week 123 - No change: number analyzed (Participants) | 20
  Week 123 - No change | 0
  Week 123 - Minimally worse: number analyzed (Participants) | 20
  Week 123 - Minimally worse | 0
  Week 123 - Much worse: number analyzed (Participants) | 20
  Week 123 - Much worse | 0
  Week 123 - Very much worse: number analyzed (Participants) | 20
  Week 123 - Very much worse | 0
  Week 135 - Very much improved: number analyzed (Participants) | 15
  Week 135 - Very much improved | 5
  Week 135 - Much improved: number analyzed (Participants) | 15
  Week 135 - Much improved | 6
  Week 135 - Minimally improved: number analyzed (Participants) | 15
  Week 135 - Minimally improved | 2
  Week 135 - No change: number analyzed (Participants) | 15
  Week 135 - No change | 1
  Week 135 - Minimally worse: number analyzed (Participants) | 15
  Week 135 - Minimally worse | 1
  Week 135 - Much worse: number analyzed (Participants) | 15
  Week 135 - Much worse | 0
  Week 135 - Very much worse: number analyzed (Participants) | 15
  Week 135 - Very much worse | 0
  Week 147 - Very much improved: number analyzed (Participants) | 7
  Week 147 - Very much improved | 4
  Week 147 - Much improved: number analyzed (Participants) | 7
  Week 147 - Much improved | 2
  Week 147 - Minimally improved: number analyzed (Participants) | 7
  Week 147 - Minimally improved | 1
  Week 147 - No change: number analyzed (Participants) | 7
  Week 147 - No change | 0
  Week 147 - Minimally worse: number analyzed (Participants) | 7
  Week 147 - Minimally worse | 0
  Week 147 - Much worse: number analyzed (Participants) | 7
  Week 147 - Much worse | 0
  Week 147 - Very much worse: number analyzed (Participants) | 7
  Week 147 - Very much worse | 0
  Week 159 - Very much improved: number analyzed (Participants) | 4
  Week 159 - Very much improved | 4
  Week 159 - Much improved: number analyzed (Participants) | 4
  Week 159 - Much improved | 0
  Week 159 - Minimally improved: number analyzed (Participants) | 4
  Week 159 - Minimally improved | 0
  Week 159 - No change: number analyzed (Participants) | 4
  Week 159 - No change | 0
  Week 159 - Minimally worse: number analyzed (Participants) | 4
  Week 159 - Minimally worse | 0
  Week 159 - Much worse: number analyzed (Participants) | 4
  Week 159 - Much worse | 0
  Week 159 - Very much worse: number analyzed (Participants) | 4
  Week 159 - Very much worse | 0
  Week 171 - Very much improved: number analyzed (Participants) | 1
  Week 171 - Very much improved | 1
  Week 171 - Much improved: number analyzed (Participants) | 1
  Week 171 - Much improved | 0
  Week 171 - Minimally improved: number analyzed (Participants) | 1
  Week 171 - Minimally improved | 0
  Week 171 - No Change: number analyzed (Participants) | 1
  Week 171 - No Change | 0
  Week 171 - Minimally worse: number analyzed (Participants) | 1
  Week 171 - Minimally worse | 0
  Week 171 - Much worse: number analyzed (Participants) | 1
  Week 171 - Much worse | 0
  Week 171 - Very much worse: number analyzed (Participants) | 1
  Week 171 - Very much worse | 0
  ET/SFU Visit - Very much improved: number analyzed (Participants) | 20
  ET/SFU Visit - Very much improved | 3
  ET/SFU Visit - Much improved: number analyzed (Participants) | 20
  ET/SFU Visit - Much improved | 8
  ET/SFU Visit - Minimally improved: number analyzed (Participants) | 20
  ET/SFU Visit - Minimally improved | 2
  ET/SFU Visit - No Change: number analyzed (Participants) | 20
  ET/SFU Visit - No Change | 4
  ET/SFU Visit - Minimally worse: number analyzed (Participants) | 20
  ET/SFU Visit - Minimally worse | 2
  ET/SFU Visit - Much worse: number analyzed (Participants) | 20
  ET/SFU Visit - Much worse | 0
  ET/SFU Visit - Very much worse: number analyzed (Participants) | 20
  ET/SFU Visit - Very much worse | 1

16. Secondary Outcome: Part B: Mean Change From Baseline in Lactate Dehydrogenase (LDH) Level at Each Specified Time Points
Description: Mean change from baseline in LDH levels at each specified time points (i.e., Weeks 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65, 67, 69, 71, 73, 75, 77, 79, 83, 87, 91, 95, 99, 103, 107, 111, 115, 119, 123, 127, 131, 135, 139, 143, 147, 151, 155, 159, 163, 167, 171, 175 and ET/SFU Visit) is reported in this outcome measure. Baseline (Week 0) was defined as the last non-missing value prior to the first administration of study drug in Part A. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 185).
Time Frame: as for outcome 9
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | BIVV009
Number analyzed (Participants) | 22
units per liter
  Week 27 | -111.59 (327.80)
  Week 29: number analyzed (Participants) | 21
  Week 29 | -129.76 (331.91)
  Week 31 | -95.27 (319.25)
  Week 33: number analyzed (Participants) | 21
  Week 33 | -82.19 (330.04)
  Week 35 | -126.64 (346.75)
  Week 37: number analyzed (Participants) | 21
  Week 37 | -151.57 (307.15)
  Week 39: number analyzed (Participants) | 15
  Week 39 | -49.27 (172.53)
  Week 41: number analyzed (Participants) | 21
  Week 41 | -116.10 (305.11)
  Week 43: number analyzed (Participants) | 19
  Week 43 | -150.26 (271.72)
  Week 45: number analyzed (Participants) | 21
  Week 45 | -85.48 (308.01)
  Week 47: number analyzed (Participants) | 21
  Week 47 | -79.81 (286.13)
  Week 49: number analyzed (Participants) | 21
  Week 49 | -104.38 (313.66)
  Week 51: number analyzed (Participants) | 19
  Week 51 | -76.84 (344.60)
  Week 53: number analyzed (Participants) | 21
  Week 53 | -87.00 (299.09)
  Week 55: number analyzed (Participants) | 21
  Week 55 | -68.29 (305.09)
  Week 57: number analyzed (Participants) | 21
  Week 57 | -101.71 (273.44)
  Week 59: number analyzed (Participants) | 21
  Week 59 | -97.71 (296.74)
  Week 61: number analyzed (Participants) | 21
  Week 61 | -89.48 (298.05)
  Week 63: number analyzed (Participants) | 20
  Week 63 | -94.20 (288.34)
  Week 65: number analyzed (Participants) | 20
  Week 65 | -91.05 (305.75)
  Week 67: number analyzed (Participants) | 19
  Week 67 | -106.32 (327.48)
  Week 69: number analyzed (Participants) | 19
  Week 69 | -75.00 (333.47)
  Week 71: number analyzed (Participants) | 18
  Week 71 | -52.39 (378.82)
  Week 73: number analyzed (Participants) | 17
  Week 73 | -70.35 (348.56)
  Week 75: number analyzed (Participants) | 19
  Week 75 | -18.68 (323.02)
  Week 77: number analyzed (Participants) | 21
  Week 77 | -64.67 (335.73)
  Week 79: number analyzed (Participants) | 20
  Week 79 | -54.10 (338.58)
  Week 83: number analyzed (Participants) | 19
  Week 83 | -87.21 (344.88)
  Week 87: number analyzed (Participants) | 18
  Week 87 | -89.17 (392.80)
  Week 91: number analyzed (Participants) | 19
  Week 91 | -78.47 (349.15)
  Week 95: number analyzed (Participants) | 16
  Week 95 | -132.75 (301.36)
  Week 99: number analyzed (Participants) | 18
  Week 99 | -13.83 (155.04)
  Week 103: number analyzed (Participants) | 20
  Week 103 | -106.40 (309.44)
  Week 107: number analyzed (Participants) | 20
  Week 107 | -85.45 (312.50)
  Week 111: number analyzed (Participants) | 19
  Week 111 | -107.58 (286.18)
  Week 115: number analyzed (Participants) | 19
  Week 115 | -107.84 (293.61)
  Week 119: number analyzed (Participants) | 19
  Week 119 | -63.68 (310.56)
  Week 123: number analyzed (Participants) | 20
  Week 123 | -58.90 (339.49)
  Week 127: number analyzed (Participants) | 18
  Week 127 | -57.72 (400.26)
  Week 131: number analyzed (Participants) | 19
  Week 131 | -113.63 (344.53)
  Week 135: number analyzed (Participants) | 17
  Week 135 | -97.06 (339.41)
  Week 139: number analyzed (Participants) | 13
  Week 139 | -1.00 (256.65)
  Week 143: number analyzed (Participants) | 10
  Week 143 | 180.70 (318.62)
  Week 147: number analyzed (Participants) | 7
  Week 147 | -10.29 (196.90)
  Week 151: number analyzed (Participants) | 8
  Week 151 | -24.13 (146.79)
  Week 155: number analyzed (Participants) | 8
  Week 155 | -17.38 (146.80)
  Week 159: number analyzed (Participants) | 4
  Week 159 | -126.00 (150.38)
  Week 163: number analyzed (Participants) | 4
  Week 163 | -31.50 (35.49)
  Week 167: number analyzed (Participants) | 2
  Week 167 | -48.50 (68.59)
  Week 171: number analyzed (Participants) | 1
  Week 171 | -23.00
  Week 175: number analyzed (Participants) | 1
  Week 175 | 6.00
  ET/SFU visit: number analyzed (Participants) | 20
  ET/SFU visit | -107.50 (249.28)

17. Secondary Outcome: Part B: Number of Blood Transfusions Per Participant
Description: A participant was to receive a transfusion if his or her Hgb level met either of the following criteria: Hgb was <9 g/dL and the participant had symptoms of anemia or Hgb was <7 g/dL and the participant was asymptomatic.
Time Frame: From Week 27 up to 149 weeks of treatment (i.e., up to Week 176)
Population: Analysis was performed on Part-B FAS. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: blood transfusions per participant
Arm/Group | BIVV009
Number analyzed (Participants) | 22
blood transfusions per participant | 2.86 (6.58)

18. Secondary Outcome: Part B: Number of Blood Units Transfused Per Participant
Description: as for outcome 17
Time Frame: From Week 27 up to 149 weeks of treatment (i.e., up to Week 176)
Population: Analysis was performed on Part B-FAS. Here, 'overall number of participants analyzed' = number of participants with at least 1 transfusion. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: blood units transfused per participants
Arm/Group | BIVV009
Number analyzed (Participants) | 7
blood units transfused per participants | 16.57 (16.85)

19. Secondary Outcome: Part B: Change From Baseline in Haptoglobin Values at Each Specified Time Points
Description: Change in Haptoglobin values from baseline at each specified time points (i.e., Weeks 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65, 67, 69, 71, 73, 75, 77, 79, 83, 87, 91, 95, 99, 103, 107, 111, 115, 119, 123, 127, 131, 135, 139, 143, 147, 151, 155, 159, 163, 167, 171, 175 and ET/SFU Visit) is reported in this outcome measure. Baseline was defined as the last non-missing value prior to the first administration of study drug in Part A. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 185). Haptoglobin values <0.2 were imputed as 0.2.
Time Frame: Baseline, Weeks 27,29,31,33,35,37,39,41,43, 45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65, 67, 69, 71, 73, 75, 77, 79, 83, 87, 91, 95, 99, 103, 107, 111, 115, 119, 123, 127, 131, 135, 139, 143, 147, 151, 155, 159, 163, 167, 171, 175, ET/SFU (up to Week 185)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | BIVV009
Number analyzed (Participants) | 22
grams per liter
  Week 27 | 0.21 (0.38)
  Week 29: number analyzed (Participants) | 21
  Week 29 | 0.21 (0.45)
  Week 31 | 0.21 (0.43)
  Week 33 | 0.28 (0.53)
  Week 35 | 0.25 (0.41)
  Week 37: number analyzed (Participants) | 21
  Week 37 | 0.14 (0.28)
  Week 39: number analyzed (Participants) | 17
  Week 39 | 0.27 (0.49)
  Week 41: number analyzed (Participants) | 20
  Week 41 | 0.39 (0.59)
  Week 43: number analyzed (Participants) | 18
  Week 43 | 0.29 (0.47)
  Week 45: number analyzed (Participants) | 21
  Week 45 | 0.16 (0.26)
  Week 47: number analyzed (Participants) | 20
  Week 47 | 0.15 (0.35)
  Week 49: number analyzed (Participants) | 21
  Week 49 | 0.21 (0.41)
  Week 51: number analyzed (Participants) | 19
  Week 51 | 0.20 (0.37)
  Week 53 | 0.23 (0.46)
  Week 55: number analyzed (Participants) | 20
  Week 55 | 0.26 (0.45)
  Week 57: number analyzed (Participants) | 20
  Week 57 | 0.26 (0.43)
  Week 59: number analyzed (Participants) | 21
  Week 59 | 0.29 (0.44)
  Week 61: number analyzed (Participants) | 21
  Week 61 | 0.23 (0.43)
  Week 63: number analyzed (Participants) | 20
  Week 63 | 0.38 (0.50)
  Week 65: number analyzed (Participants) | 20
  Week 65 | 0.25 (0.41)
  Week 67: number analyzed (Participants) | 19
  Week 67 | 0.25 (0.42)
  Week 69: number analyzed (Participants) | 20
  Week 69 | 0.24 (0.47)
  Week 71: number analyzed (Participants) | 19
  Week 71 | 0.19 (0.33)
  Week 73: number analyzed (Participants) | 19
  Week 73 | 0.13 (0.29)
  Week 75: number analyzed (Participants) | 20
  Week 75 | 0.13 (0.24)
  Week 77: number analyzed (Participants) | 21
  Week 77 | 0.17 (0.29)
  Week 79: number analyzed (Participants) | 20
  Week 79 | 0.09 (0.22)
  Week 83: number analyzed (Participants) | 20
  Week 83 | 0.14 (0.25)
  Week 87: number analyzed (Participants) | 18
  Week 87 | 0.35 (0.53)
  Week 91: number analyzed (Participants) | 19
  Week 91 | 0.17 (0.28)
  Week 95: number analyzed (Participants) | 20
  Week 95 | 0.19 (0.33)
  Week 99: number analyzed (Participants) | 18
  Week 99 | 0.21 (0.37)
  Week 103: number analyzed (Participants) | 21
  Week 103 | 0.15 (0.25)
  Week 107: number analyzed (Participants) | 21
  Week 107 | 0.26 (0.40)
  Week 111: number analyzed (Participants) | 19
  Week 111 | 0.22 (0.33)
  Week 115: number analyzed (Participants) | 18
  Week 115 | 0.21 (0.35)
  Week 119: number analyzed (Participants) | 19
  Week 119 | 0.16 (0.31)
  Week 123: number analyzed (Participants) | 20
  Week 123 | 0.19 (0.45)
  Week 127: number analyzed (Participants) | 20
  Week 127 | 0.14 (0.23)
  Week 131: number analyzed (Participants) | 19
  Week 131 | 0.18 (0.38)
  Week 135: number analyzed (Participants) | 18
  Week 135 | 0.18 (0.35)
  Week 139: number analyzed (Participants) | 13
  Week 139 | 0.10 (0.17)
  Week 143: number analyzed (Participants) | 11
  Week 143 | 0.07 (0.16)
  Week 147: number analyzed (Participants) | 8
  Week 147 | 0.06 (0.16)
  Week 151: number analyzed (Participants) | 8
  Week 151 | 0.12 (0.24)
  Week 155: number analyzed (Participants) | 8
  Week 155 | 0.09 (0.22)
  Week 159: number analyzed (Participants) | 5
  Week 159 | 0.15 (0.34)
  Week 163: number analyzed (Participants) | 4
  Week 163 | 0.30 (0.35)
  Week 167: number analyzed (Participants) | 2
  Week 167 | 0.00 (0.00)
  Week 171: number analyzed (Participants) | 1
  Week 171 | 0.00
  Week 175: number analyzed (Participants) | 1
  Week 175 | 0.00
  ET/SFU visit: number analyzed (Participants) | 20
  ET/SFU visit | 0.02 (0.13)

20. Secondary Outcome: Part B: Number of Healthcare Visits by Type
Description: In this outcome measure, number of healthcare visits which included non-study healthcare resource utilization visit (consisted mainly of extra visits to the office of the study doctor, or visit to a generalist doctor, or visit to a specialist doctor) and hospitalization visit and visit to hospital emergency is reported.
Time Frame: From Week 27 up to 149 weeks of treatment (i.e., up to Week 176)
Population: Analysis was performed on Part B-FAS. Data for this outcome measure was planned to be collected and analyzed for combined population (i.e., all participants who received BIVV009 [either at 6.5 g or 7.5 g]).
Measure: Number; unit: visits
Arm/Group | BIVV009
Number analyzed (Participants) | 22
visits
  Non-study healthcare resource utilization visits | 16
  Hospitalization | 8
  Visit to a hospital emergency room | 3

ADVERSE EVENTS:
Time Frame: Part A (both 6.5 g and 7.5 g cohorts): From first dose (Day 0) up to Week 26; Part B, 6.5 g cohort: From first dose (Week 27) up to 143 weeks of treatment + 9 weeks of follow-up (i.e., up to Week 179). Part B, 7.5 g cohort: From first dose (Week 27) up to 149 weeks of treatment + 9 weeks of follow-up (i.e., up to Week 185)
Description: Reported AEs and SAEs including fatal AEs were TEAEs that developed/worsened or became serious during on-treatment period. Analysis was performed on SAS.
Groups:
- Part A: BIVV009 6.5 g: Participants with primary CAD and body weight <75 kg with a recent history of blood transfusion (defined as at least 1 transfusion during the last 6 months prior to screening in this study) received an IV infusion of BIVV009 6.5 g on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25.
- Part A: BIVV009 7.5 g: Participants with primary CAD and body weight >=75 kg with a recent history of blood transfusion (defined as at least 1 transfusion during the last 6 months prior to screening in this study) received an IV infusion of BIVV009 7.5 g on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25.
- Part B: BIVV009 6.5 g: Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 6.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 143 weeks. All participants who completed Part A elected to continue in Part B.
- Part B: BIVV009 7.5 g: Participants who completed Part A per protocol through the end of treatment visit (Week 26) could continue to receive BIVV009 7.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 149 weeks. All participants who completed Part A elected to continue in Part B.
Arm/Group | Part A: BIVV009 6.5 g | Part A: BIVV009 7.5 g | Part B: BIVV009 6.5 g | Part B: BIVV009 7.5 g
All-Cause Mortality (participants affected / at risk) | 0/17 | 1/7 | 2/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/17 | 3/7 | 10/16 | 2/6
Other Adverse Events (participants affected / at risk) | 15/17 | 6/7 | 16/16 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: BIVV009 6.5 g (N=17) | Part A: BIVV009 7.5 g (N=7) | Part B: BIVV009 6.5 g (N=16) | Part B: BIVV009 7.5 g (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold Type Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asymptomatic Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumococcal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound Infection Staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tubular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient Global Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyanosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Peripheral Artery Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: BIVV009 6.5 g (N=17) | Part A: BIVV009 7.5 g (N=7) | Part B: BIVV009 6.5 g (N=16) | Part B: BIVV009 7.5 g (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 5 (11) | 2 (2)
Cold Type Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monoclonal B-Cell Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic Valve Sclerosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tricuspid Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniere's Disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular Degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular Discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Field Defect (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (8)
Abdominal Tenderness (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (5)
Oral Mucosal Blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (4) | 1 (1)
Catheter Site Haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device Related Thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (5)
Feeling Cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (2)
Peripheral Swelling (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (4)
Temperature Intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Allergy To Arthropod Bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoinflammatory Disease (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asymptomatic Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (7) | 1 (1)
Cystitis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (3) | 0 (0)
Herpes Simplex Viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 4 (6) | 0 (0)
Oral Herpes (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Otitis Externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis Externa Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Root Canal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea Pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (4) | 0 (0) | 1 (1) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (13) | 2 (6)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Exposure To Extreme Temperature (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 1 (1) | 1 (1) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal Column Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Immunoglobulin G Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-Reactive Protein Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest X-Ray Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Computerised Tomogram Head Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum Ferritin Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Magnesium Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral Disc Calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain Oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Dizziness Postural (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adjustment Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental Fatigue (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 0 (0) | 2 (6) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restrictive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodular Vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Air Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory Collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyanosis (Vascular disorders) | 2 (3) | 0 (0) | 2 (3) | 2 (4)
Essential Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibromuscular Dysplasia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 3 (6) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT03347396/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03347396/SAP_001.pdf